CLINICAL TRIAL: NCT04010955
Title: The Role of Additional Antiplatelet Therapy in the Ischemic Stroke With Atrial Fibrillation and Co-morbiD Atherosclerosis During edOxaban treatmeNt. (ADD-ON) Study, Multicenter Registry-based Analysis
Brief Title: Adding Antiplatelet During Edoxaban Treatment in Stroke Patients With Non-valvular Atrial Fibrillation (ADD-ON)
Acronym: (ADD-ON)
Status: Active, not recruiting | Type: Observational
Sponsor: Asan Medical Center (Other)
Collaborators: Samsung Medical Center (Other); Myongji Hospital (Other); Ewha Womans University (Other); Chonbuk National University (Other); Pusan National University Hospital (Other); Korea University Ansan Hospital (Other); Keimyung University Dongsan Medical Center (Other); Chonnam National University Hospital (Other); Korea University Guro Hospital (Other); Chungnam National University Hospital (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Kyungpook National University Hospital (Other); Dongtan Sacred Heart Hospital (Other); Eulji University Hospital (Other)
Responsible Party: Principal Investigator, Sun U. Kwon, Professor, Asan Medical Center
Other Study IDs: Add-on_001
Record Dates: First submitted 2019-06-24; First posted 2019-07-08 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-07

CONDITIONS: Acute Ischemic Stroke; Atrial Fibrillation; Extracranial Atherosclerosis; Intracranial Atherosclerosis; Coronary Artery Atherosclerosis; Peripheral Artery Stenosis; Anticoagulant; Antiplatelet
MeSH Terms: conditions — Ischemic Stroke; Atrial Fibrillation; Intracranial Arteriosclerosis; Coronary Artery Disease | interventions — edoxaban

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Edoxaban Monotherapy: edoxaban monotherapy without additional antiplatelet therapy in long term stroke prevention.
  However, transient additional antiplatelet therapy will be allowed at the discretion of duty physicians.
  Interventions: Drug: Edoxaban Monotherapy
- Edoxaban and antiplatelet combination: edoxaban plus additional antiplatelet therapy in long term stroke prevention. However, transient cessation of antiplatelet therapy will be allowed at the discretion of duty physicians.
  Interventions: Drug: Edoxaban Monotherapy

INTERVENTIONS:
Drug: Edoxaban Monotherapy — when the patients will be initially registered in this study, duty physicians will make a decision to give additional antiplatelet therapy in addition to standard edoxaban therapy.
  Other Names: Edoxaban and antiplatelet combination

SUMMARY:
This study aims to compare the effectiveness and safety regarding treatment with standard anticoagulant only or adding antiplatelet to anticoagulant in patients with non-valvular atrial fibrillation and significant atherosclerosis including extracranial, intracranial, coronary or peripheral artery.

DETAILED DESCRIPTION:
Although there is a significant increase in the risk of cerebral infarction in the presence of atrial fibrillation, it is difficult to say that all cerebral infarctions occurring in patients with atrial fibrillation are caused by atrial fibrillation. Carotid stenosis is found in 1/4 of patients with atrial fibrillation, which increases the risk of cerebral infarction. Additional antiplatelet therapy to standard anticoagulation therapy should be considered in some patients. To date, the best medical treatment for prevention of cerebral infarction in patients with atrial fibrillation and accompanying atherosclerosis has not been evaluated yet.

Edoxaban reduced bleeding complication compared to warfarin in patients with atrial fibrillation. In addition, the ENGAGE AF TIMI-48 study showed a tendency to reduce cerebral infarction (p for interaction = 0.08) when administered in combination with one antiplatelet agent and edoxaban. The administration of antiplatelet agents may be due to patients had accompanying myocardial infarction or cerebral infarction. This group is also thought to have a high risk of bleeding due to high HAS-BLED scores. Nonetheless, there was a similar degree of bleeding in patients receiving additional antiplatelet agents. There was also less bleeding in the warfarin arm than in the use of additional antiplatelet agents. (Major bleeding: 0.19 vs 0.24% / yr; intracranial hemorrhage: 0.43 vs 0.57% / yr)

Thus, Edoxaban have good clinical trial results in combination with antiplatelet agents in atrial fibrillation with atherosclerosis compared to other NOACs(new oral anticoagulants). It is also considered to be suitable for combination therapy with antiplatelet agents because of its advantages in different bleeding compared to other warfarin. However, there is no evidence to suggest that Edoxaban alone or in combination with additional antiplatelet agents is better for stroke patients with atrial fibrillation and significant arteriosclerosis.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with acute cerebral infarction or transient ischemic attack within 14 days of symptom onset based on Last Known Normal Time.
2. Patients with non-valvular atrial fibrillation including paroxysmal atrial fibrillation which is eligible for treatment with Edoxaban.
3. Patients with significant atherosclerosis confirmed by imaging tests on the cerebral arteries, coronary arteries, or peripheral arteries and suitable for the use of antiplatelet agents.

   * Significant intracranial internal stenosis confirmed by CTA or MRA
   * A history of coronary artery disease, meaningful findings from CTA or CAG Arterial stenosis
   * Peripheral arterial disease (Ankle-Brachial Index, ABI <0.9, significant stenosis found in lower limb ultrasonography

3) Men and women over 20 years old 4) Patients who voluntarily agreed to register the registry

Exclusion Criteria:

1. Patients with chronic renal failure (GFR <30 ml / min) or severe liver damage
2. patients requiring warfarin medication due to prosthetic valve replacement
3. patients with internal bleeding (active internal bleeding)
4. bleeding diathesis
5. History of acute myocardial infarction or received coronary artery procedure within 6 months before screening
6. Patients who have received or are scheduled to undergo carotid stenting within 1 year
7. Currently, two or more antiplatelet agents are required due to arteriosclerosis.
8. Patients whose survival period is expected to be less than 12 months due to serious diseases such as terminal cancer or liver failure
9. Patients who are scheduled for invasive surgery with possible uncontrolled bleeding, including major surgery
10. Women who are pregnant or lactating, do not have contraception during the study
11. A person who is found to be unsuitable for participation in the study due to the clinical laboratory test results or other reasons

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with acute cerebral infarction or transient ischemic attack with non-valvular atrial fibrillation and significant artherosclerosis
  Significant atherosclerosis means atherosclerosis in the cerebral, coronary or peripheral arteries according to the judgment of the researchers.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2019-10-08 (Actual); Primary Completion 2025-06-27 (Actual); Study Completion 2026-06-27 (Estimated)

PRIMARY OUTCOMES:
MACE (major adverse cardiac event) | 18 months
  Duration for first occurrence of major cardiovascular events after patient registration: ischemic stroke, hemorrhagic stroke, myocardial infarction, vascular death

SECONDARY OUTCOMES:
Hemorrhagic stroke | 18 months
  Duration for first occurrence of hemorrhagic stroke after patient registration
Stroke | 18 months
  Duration for first occurrence of stroke (ischemic and hemorrhagic) after patient registration
Acute Myocardial Infarction | 18 months
  Duration for first occurrence of acute myocardial infarction after patient registration
Major bleeding | 18 months
  Duration for occurrence of major bleeding based on ISTH( International Society on Thrombosis and Haemostasis) after patient registration
Vascular death | 18 months
  Duration for first occurrence of vascular death after patient registration
Ischemic stroke | 18 months
  Duration for first occurrence of ischemic stroke after patient registration
Net clinical benefit based on reduction in major adverse cardiac event compared to major bleeding events | 18 months
  Net clinical benefit based on reduction in major adverse cardiac event compared to major bleeding events

CONTACTS AND LOCATIONS:
Overall Officials: Sun U. Kwon, MD, PhD, Principal Investigator — Asan Medical Center
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Ogilvie IM, Newton N, Welner SA, Cowell W, Lip GY. Underuse of oral anticoagulants in atrial fibrillation: a systematic review. Am J Med. 2010 Jul;123(7):638-645.e4. doi: 10.1016/j.amjmed.2009.11.025. PMID 20609686
- [Background] Willeit K, Pechlaner R, Egger G, Weger S, Oberhollenzer M, Willeit J, Kiechl S. Carotid atherosclerosis and incident atrial fibrillation. Arterioscler Thromb Vasc Biol. 2013 Nov;33(11):2660-5. doi: 10.1161/ATVBAHA.113.302272. Epub 2013 Sep 12. PMID 24030550
- [Background] Kanter MC, Tegeler CH, Pearce LA, Weinberger J, Feinberg WM, Anderson DC, Gomez CR, Rothrock JF, Helgason CM, Hart RG. Carotid stenosis in patients with atrial fibrillation. Prevalence, risk factors, and relationship to stroke in the Stroke Prevention in Atrial Fibrillation Study. Arch Intern Med. 1994 Jun 27;154(12):1372-7. PMID 8002689
- [Background] Chang YJ, Ryu SJ, Lin SK. Carotid artery stenosis in ischemic stroke patients with nonvalvular atrial fibrillation. Cerebrovasc Dis. 2002;13(1):16-20. doi: 10.1159/000047740. PMID 11810005
- [Background] Lehtola H, Airaksinen KEJ, Hartikainen P, Hartikainen JEK, Palomaki A, Nuotio I, Ylitalo A, Kiviniemi T, Mustonen P. Stroke recurrence in patients with atrial fibrillation: concomitant carotid artery stenosis doubles the risk. Eur J Neurol. 2017 May;24(5):719-725. doi: 10.1111/ene.13280. Epub 2017 Mar 20. PMID 28317289
- [Background] Hart RG, Pearce LA, Aguilar MI. Meta-analysis: antithrombotic therapy to prevent stroke in patients who have nonvalvular atrial fibrillation. Ann Intern Med. 2007 Jun 19;146(12):857-67. doi: 10.7326/0003-4819-146-12-200706190-00007. PMID 17577005
- [Background] Chimowitz MI, Lynn MJ, Howlett-Smith H, Stern BJ, Hertzberg VS, Frankel MR, Levine SR, Chaturvedi S, Kasner SE, Benesch CG, Sila CA, Jovin TG, Romano JG; Warfarin-Aspirin Symptomatic Intracranial Disease Trial Investigators. Comparison of warfarin and aspirin for symptomatic intracranial arterial stenosis. N Engl J Med. 2005 Mar 31;352(13):1305-16. doi: 10.1056/NEJMoa043033. PMID 15800226
- [Background] Fisher M. Does the combination of warfarin and aspirin have a place in secondary stroke prevention? No. Stroke. 2009 May;40(5):1944-5. doi: 10.1161/STROKEAHA.108.537670. Epub 2009 Mar 19. No abstract available. PMID 19299634
- [Background] Kim BJ, Kim HJ, Do Y, Lee JH, Park KY, Cha JK, Kim HY, Kwon JH, Lee KB, Kim DE, Ha SW, Sohn SI, Kwon SU. The impact of prior antithrombotic status on cerebral infarction in patients with atrial fibrillation. J Stroke Cerebrovasc Dis. 2014 Sep;23(8):2054-2059. doi: 10.1016/j.jstrokecerebrovasdis.2014.03.011. Epub 2014 Aug 10. PMID 25113085
- [Background] Connolly SJ, Ezekowitz MD, Yusuf S, Eikelboom J, Oldgren J, Parekh A, Pogue J, Reilly PA, Themeles E, Varrone J, Wang S, Alings M, Xavier D, Zhu J, Diaz R, Lewis BS, Darius H, Diener HC, Joyner CD, Wallentin L; RE-LY Steering Committee and Investigators. Dabigatran versus warfarin in patients with atrial fibrillation. N Engl J Med. 2009 Sep 17;361(12):1139-51. doi: 10.1056/NEJMoa0905561. Epub 2009 Aug 30. PMID 19717844
- [Background] Kim BJ, Kang HG, Lee DH, Kang DW, Kim JS, Kwon SU. Ischemic stroke on optimal anticoagulation with novel-oral anticoagulants compared with warfarin. Int J Stroke. 2015 Aug;10(6):E68. doi: 10.1111/ijs.12587. No abstract available. PMID 26202718
- [Background] Giugliano RP, Ruff CT, Braunwald E, Murphy SA, Wiviott SD, Halperin JL, Waldo AL, Ezekowitz MD, Weitz JI, Spinar J, Ruzyllo W, Ruda M, Koretsune Y, Betcher J, Shi M, Grip LT, Patel SP, Patel I, Hanyok JJ, Mercuri M, Antman EM; ENGAGE AF-TIMI 48 Investigators. Edoxaban versus warfarin in patients with atrial fibrillation. N Engl J Med. 2013 Nov 28;369(22):2093-104. doi: 10.1056/NEJMoa1310907. Epub 2013 Nov 19. PMID 24251359
- [Background] Perez-Gomez F, Alegria E, Berjon J, Iriarte JA, Zumalde J, Salvador A, Mataix L; NASPEAF Investigators. Comparative effects of antiplatelet, anticoagulant, or combined therapy in patients with valvular and nonvalvular atrial fibrillation: a randomized multicenter study. J Am Coll Cardiol. 2004 Oct 19;44(8):1557-66. doi: 10.1016/j.jacc.2004.05.084. PMID 15489085
- [Background] Ois A, Cuadrado-Godia E, Rodriguez-Campello A, Giralt-Steinhauer E, Jimenez-Conde J, Lopez-Cuina M, Ley M, Soriano C, Roquer J. Relevance of stroke subtype in vascular risk prediction. Neurology. 2013 Aug 6;81(6):575-80. doi: 10.1212/WNL.0b013e31829e6f37. Epub 2013 Jul 3. PMID 23825174
- [Background] Kang K, Park TH, Kim N, Jang MU, Park SS, Park JM, Ko Y, Lee S, Lee KB, Lee J, Kim DE, Cho YJ, Kim JT, Kim DH, Cha JK, Han MK, Lee JS, Lee J, Oh MS, Choi JC, Lee BC, Hong KS, Bae HJ. Recurrent Stroke, Myocardial Infarction, and Major Vascular Events during the First Year after Acute Ischemic Stroke: The Multicenter Prospective Observational Study about Recurrence and Its Determinants after Acute Ischemic Stroke I. J Stroke Cerebrovasc Dis. 2016 Mar;25(3):656-64. doi: 10.1016/j.jstrokecerebrovasdis.2015.11.036. Epub 2015 Dec 29. PMID 26750575